CLINICAL TRIAL: NCT03570619
Title: IMPACT: Immunotherapy in Patients With Metastatic Cancers and CDK12 Mutations
Brief Title: Immunotherapy in Patients With Metastatic Cancers and CDK12 Mutations
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.050; HUM00145104 (Other: University of Michigan)
Record Dates: First submitted 2018-06-15; First posted 2018-06-27 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer; Metastatic Cancer; Solid Tumor
Keywords: Metastatic Cancer; Metastatic Castration Resistant Prostate Cancer; mCRPC; Immunotherapy; CDK12; Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Metastatic CRPC (Experimental): Patients with metastatic castration resistant prostate cancer (mCRPC) will be enrolled in cohort A.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Solid Tumors (non-prostate) (Experimental): Patients with all other metastatic subtypes will be enrolled in cohort B
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Metastatic CRPC with Monotherapy (Experimental): Patients with metastatic castration resistant prostate cancer (mCRPC) will be enrolled in cohort C once enrollment to cohort A has been completed.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Patients in arms Metastatic CRPC and Experimental: Solid Tumors (non-prostate) will begin receiving combination therapy with nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV every 3 weeks for up to 4 cycles if tolerated, followed by nivolumab maintenance therapy at flat dose 480 mg IV every 4 weeks through the end of the planned study duration, for up to 104 weeks of total therapy.
  Patients in arm Metastatic CRPC will receive therapy with monotherapy nivolumab therapy at flat dose 480 mg IV every 4 weeks for up to 104 weeks of total therapy.
Drug: Ipilimumab — Patients in arms Metastatic CRPC and Experimental: Solid Tumors (non-prostate) will begin receiving combination therapy with nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV every 3 weeks for up to 4 cycles if tolerated, followed by nivolumab maintenance therapy at flat dose 480 mg IV every 4 weeks through the end of the planned study duration, for up to 104 weeks of total therapy.
  Arms: Metastatic CRPC; Solid Tumors (non-prostate)

SUMMARY:
This study will attempt to determine the efficacy of checkpoint inhibitor immunotherapy with nivolumab and ipilimumab combination therapy followed by nivolumab monotherapy in patients with metastatic prostate cancer and other tumor solid tumor histologies harboring loss of CDK12 function as well as monotherapy nivolumab treatment in patient with metastatic prostate cancer harboring loss of CDK12 function.

DETAILED DESCRIPTION:
This study investigates the efficacy of checkpoint inhibitor immunotherapy in patients with metastatic cancer with CDK12 mutations. The study includes three cohorts: Cohort A consists of metastatic prostate cancer patients being treated with combination nivolumab and ipilimumab treatment followed by monotherapy nivolumab treatment. Cohort B consists of other solid tumor patients being treated with combination nivolumab and ipilimumab treatment followed by monotherapy nivolumab treatment. As of an amendment approved 03FEB2021 a third cohort was added, Cohort C, which consists of metastatic prostate cancer patients being treated with monotherapy nivolumab treatment.

As of an amendment approved 21JUN2020 the maximum duration of treatment, as well as the anticipated timing for some of the studies outcome measures, were updated from 52 weeks to 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age as of date of signing informed consent.
* Be willing and able to provide written informed consent for the study.
* ECOG Performance Status of 0, 1 or 2 (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death.
* Subjects must have a histologic or cytologic diagnosis of metastatic adenocarcinoma of the prostate without small cell histology OR another type of metastatic carcinoma.
* All subjects, regardless of cancer type, must have a documented CDK12 aberration in tumor tissue.
* Subjects with prostate cancer must have documented prostate cancer progression within six months prior to screening with PSA progression defined as a minimum of three rising PSA levels ≥ 1; 1 week between each assessment with a baseline PSA value at screening of ≥ 2 ng/mL.
* Subjects with prostate cancer must have ongoing androgen deprivation with total serum testosterone < 50 ng/dL (or ≤ 0.50 ng/mL or 1.73 nmol/L)). If the subject is currently being treated with LHRH agonists (subjects who have not undergone an orchiectomy), this therapy must have been initiated at least 4 weeks prior to registration. This treatment must be continued throughout the study.
* Subjects with non-prostate histologies must have RECIST 1.1-measurable cancer on computed tomography (CT) or magnetic resonance imaging (MRI) scans.
* Subjects must have recovered to baseline or ≤ grade 1 toxicities related to any prior treatments unless AE(s) are clinically non-significant and/or stable.
* Patients must be ≥ 2 weeks from most recent systemic therapy or most recent radiation therapy.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 28 days prior to registration.
* Female and male subjects of reproductive potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 5 months (for women) and 7 months (for men) after the last dose of study therapy.
* Adequate organ and marrow function

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1 and anti-CTLA-4 is NOT allowed. Prior intravesical BCG therapy is allowed.
* Treatment with any investigational agent or on an interventional clinical trial within 28 days prior to registration.
* Prior or concurrent malignancy except for: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, localized or locally advanced prostate cancer definitively treated without recurrence or with biochemical recurrence only, or any other cancer fully treated or from which the subject has been disease-free for at least 2 years.
* Autoimmune diseases such as rheumatoid arthritis. Vitiligo, mild psoriasis (topical therapy only) or hypothyroidism are allowed.
* Need for systemic corticosteroids >10mg prednisone daily or equivalent alternative steroid (except physiologic dose for adrenal replacement therapy) or other immunosuppressive agents (such as cyclosporine or methotrexate) Topical and inhaled corticosteroids are allowed if medically needed.
* Any history of organ allografts
* Any history of HIV, hepatitis B or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, MD, Principal Investigator — Rogel Cancer Center
Locations (8):
- United States (8):
  - University of California San Diego, Moores Cancer Center, San Diego, California
  - University of California San Francisco/Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - H. Lee. Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic CRPC: Patients with metastatic castration resistant prostate cancer (mCRPC) will be enrolled in cohort A.
  Nivolumab: Patients in arms Metastatic CRPC and Experimental: Solid Tumors (non-prostate) will begin receiving combination therapy with nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV every 3 weeks for up to 4 cycles if tolerated, followed by nivolumab maintenance therapy at flat dose 480 mg IV every 4 weeks through the end of the planned study duration, for up to 104 weeks of total therapy.
  Patients in arm Metastatic CRPC will receive therapy with monotherapy nivolumab therapy at flat dose 480 mg IV every 4 weeks for up to 104 weeks of total therapy.
  Ipilimumab: Patients in arms Metastatic CRPC and Experimental: Solid Tumors (non-prostate) will begin receiving combination therapy with nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV every 3 weeks for up to 4 cycles if tolerated, followed by nivolumab maintenance therapy at flat dose 480 mg IV every 4 weeks through the end of the planned study duration, for up to 104 weeks of total therapy.
- Solid Tumors (Non-prostate): Patients with all other metastatic subtypes will be enrolled in cohort B
  Nivolumab: Patients in arms Metastatic CRPC and Experimental: Solid Tumors (non-prostate) will begin receiving combination therapy with nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV every 3 weeks for up to 4 cycles if tolerated, followed by nivolumab maintenance therapy at flat dose 480 mg IV every 4 weeks through the end of the planned study duration, for up to 104 weeks of total therapy.
  Patients in arm Metastatic CRPC will receive therapy with monotherapy nivolumab therapy at flat dose 480 mg IV every 4 weeks for up to 104 weeks of total therapy.
  Ipilimumab: Patients in arms Metastatic CRPC and Experimental: Solid Tumors (non-prostate) will begin receiving combination therapy with nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV every 3 weeks for up to 4 cycles if tolerated, followed by nivolumab maintenance therapy at flat dose 480 mg IV every 4 weeks through the end of the planned study duration, for up to 104 weeks of total therapy.
- Metastatic CRPC With Monotherapy: Patients with metastatic castration resistant prostate cancer (mCRPC) will be enrolled in cohort C once enrollment to cohort A has been completed.
  Nivolumab: Patients in arms Metastatic CRPC and Experimental: Solid Tumors (non-prostate) will begin receiving combination therapy with nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV every 3 weeks for up to 4 cycles if tolerated, followed by nivolumab maintenance therapy at flat dose 480 mg IV every 4 weeks through the end of the planned study duration, for up to 104 weeks of total therapy.
  Patients in arm Metastatic CRPC will receive therapy with monotherapy nivolumab therapy at flat dose 480 mg IV every 4 weeks for up to 104 weeks of total therapy.
Period: Overall Study
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Started | 33 | 8 | 15
Completed | 29 | 5 | 14
Not Completed | 4 | 3 | 1
Not completed — Adverse Event | 2 | 0 | 1
Not completed — new diagnosis of new malignancy | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy | Total
Number analyzed (Participants) | 33 | 8 | 15 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 7 | 21
  >=65 years | 25 | 2 | 8 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 0 | 8
  Male | 33 | 0 | 15 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 31 | 8 | 15 | 54
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 0 | 2 | 8
  White | 25 | 8 | 12 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 8 | 15 | 56

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With CDK12 Loss of Function Metastatic CRPC That Respond to Treatment.
Description: The primary objective is overall response rate (ORR) of patients with metastatic CRPC. Response will be defined as a 50% decline in PSA (prostate specific antigen) from baseline as determined by PCWG3 criteria.
Time Frame: Up to 24 months post treatment
Population: only subjects who received at least 1 cycle(s) of therapy, and who have 2 PSA measurements after protocol therapy initiation were considered evaluable for PSA response.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 23 | 0 | 14
participants | 2 [1 to 28] |  | 0 [0 to 0]

2. Secondary Outcome: The Proportion of Patients That Respond to Treatment in Cohort B.
Description: Overall response will be defined as patients that achieve either a partial response or complete response using RECIST 1.1 criteria.
  Complete response (CR) is defined as disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
  Partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
Time Frame: Up to 104 weeks after start of therapy
Population: Only Cohort B analyzed and only 3 patients were evaluable per RECIST
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 0 | 3 | 0
Participants | 0 | 1 | 0

3. Secondary Outcome: Radiographic Progression Free Survival Time (rPFS)
Description: Radiographic progression-free survival (rPFS) is defined as the duration of time from start of treatment to time of radiographic progression. Progression is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: Up to 104 weeks after start of therapy
Population: numbers updated to include only evaluable patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 15 | 3 | 3
days | 166 [92 to 338] | NA [82 to NA] — NA estimates indicate not reached | 110 [92 to NA] — NA estimates indicate not reached

4. Secondary Outcome: Progression Free Survival Time (PFS)
Description: Progression is defined as the duration of time from start of treatment to time of progression. Progression is defined as:
  Either, Radiographic progression: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions OR, PSA Progression: For rising PSA after an initial decline from baseline, the PSA is recorded from the start of therapy to first PSA increase that is ≥ 25% and ≥ 2ng/mL above the nadir, which is confirmed by a second value 4 or more weeks later, confirming a rising trend. If there is no initial decline from baseline, PSA progression is defined as ≥ 25% increase and ≥ 2 ng/mL increase from baseline beyond 12 weeks.
Time Frame: Up to 24 months post treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 23 | 3 | 14
days | 213 [110 to 346] | NA [82 to NA] — NA estimates indicate not reached | 138 [105 to 421]

5. Secondary Outcome: Duration of Therapy (DOT)
Description: Defined by the time interval from the start of treatment to the day of permanent discontinuation of treatment (including death).
Time Frame: Up to 104 weeks after start of therapy
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 33 | 8 | 15
weeks | 12 [9.79 to 18.36] | 8.07 [5.71 to 19.29] | 15.86 [12.14 to 29.14]

6. Secondary Outcome: Progression Rate at 6 Months
Description: Progression is defined as: Either, Radiographic progression: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions OR, PSA Progression: For rising PSA after an initial decline from baseline, the PSA is recorded from the start of therapy to first PSA increase that is ≥ 25% and ≥ 2ng/mL above the nadir, which is confirmed by a second value 4 or more weeks later, confirming a rising trend. If there is no initial decline from baseline, PSA progression is defined as ≥ 25% increase and ≥ 2 ng/mL increase from baseline beyond 12 weeks.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 33 | 3 | 15
percentage of Participants | 74 [54 to 87] | 67 [21 to 94] | 71 [45 to 88]

7. Secondary Outcome: Overall Survival Time
Description: Defined as the time from the start of treatment until death from any cause. Patients alive or lost to follow-up at the time of analysis will be censored at their last date of follow-up.
Time Frame: Up to 24 months post treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 32 | 8 | 15
days | 273 [190 to 375] | NA [191 to NA] — NA estimates indicate not reached | 421 [111 to NA] — NA estimates indicate not reached

8. Secondary Outcome: PSA Progression Free Survival Time
Description: PSA Progression: For rising PSA after an initial decline from baseline, the PSA is recorded from the start of therapy to first PSA increase that is ≥ 25% and ≥ 2ng/mL above the nadir, which is confirmed by a second value 4 or more weeks later, confirming a rising trend. If there is no initial decline from baseline, PSA progression is defined as ≥ 25% increase and ≥ 2 ng/mL increase from baseline beyond 12 weeks.
Time Frame: Up to 24 months post treatment
Population: Only evaluable prostate cancer patients were analyzed as PSA is only collected for prostate cancer participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 23 | 0 | 14
days | 213 [110 to 346] |  | 138 [105 to 421]

9. Secondary Outcome: Time to PSA Progression
Description: as for outcome 8
Time Frame: Up to 24 months post treatment
Population: Only evaluable prostate cancer patients were analyzed as PSA is only collected for prostate cancer participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
Number analyzed (Participants) | 23 | 0 | 14
days | NA [149 to NA] — NA estimates indicate not reached |  | NA [116 to NA] — NA estimates indicate not reached

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 100 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 100 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 4.5 year period. An average of 6.5 months per participant.
Arm/Group | Metastatic CRPC | Solid Tumors (Non-prostate) | Metastatic CRPC With Monotherapy
All-Cause Mortality (participants affected / at risk) | 21/33 | 3/8 | 6/15
Serious Adverse Events (participants affected / at risk) | 16/33 | 6/8 | 4/15
Other Adverse Events (participants affected / at risk) | 32/33 | 7/8 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic CRPC (N=33) | Solid Tumors (Non-prostate) (N=8) | Metastatic CRPC With Monotherapy (N=15)
Abdominal distension (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (General disorders) | 1 (2) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Anorexia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Bacteremia
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — acute myeloid leukemia
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — immune mediated hepatitis
Hoarseness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 1 (1) — disease progression
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Cord compression
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (General disorders) | 1 (1) | 1 (1) | 0 (0)
Paroxysmal atrial tachycardia (Vascular disorders) | 1 (1) | 0 (0) | 0
Pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (General disorders) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic CRPC (N=33) | Solid Tumors (Non-prostate) (N=8) | Metastatic CRPC With Monotherapy (N=15)
Abdominal Pain (General disorders) | 2 (4) | 2 (3) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Anemia (Investigations) | 5 (10) | 1 (1) | 5 (8)
Anorexia (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 6 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 3 (3) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 4 (4) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (12) | 2 (2) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (3)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 3 (6)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 2 (3) | 5 (6)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3) | 3 (3)
Edema limbs (General disorders) | 4 (4) | 0 (0) | 2 (4)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 2 (4)
Fatigue (General disorders) | 15 (20) | 2 (2) | 7 (8)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (3) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9) | 2 (3) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 8 (9) | 0 (0) | 0 (0)
Pain in extremity (General disorders) | 2 (3) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 1 (2)
Pulmonary hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2) | 3 (4)
Weight loss (Investigations) | 3 (5) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Localized edema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (General disorders) | 0 (0) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other sites/PI's are not to publish

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03570619/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03570619/ICF_001.pdf